CLINICAL TRIAL: NCT05715177
Title: Influence of Kinesio Tapping on Quadriceps Muscle Peak Torque and Bioelectrical Activity After Arthroscopic Partial Meniscectomy (RTC)
Brief Title: Influence of Kinesio Tapping on Quadriceps Muscle Peak Torque and Bioelectrical Activity After Meniscectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Mohamed Moustafa Mohamed Ahmed, Assistant profosser of Biomechanics faculty of applied medical sciences, Jazan University KSA., University of Jazan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1147
Record Dates: First submitted 2022-12-16; First posted 2023-02-06 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Meniscus Tear

STUDY DESIGN:
Intervention Model Description: A Pretest post-test control group design will be used to investigate the effect of kinesio-taping on electrical activity and peak torque of the quadriceps femoris muscle during concentric and eccentric contraction after arthroscopic partial meniscectomy (APM) surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cura kinesio-taping (Experimental): consisted of 25 subjects who will receive kinesio-taping from origin to insertion on the superficial muscles of Quadriceps femoris (QF) (Vastus Medialis (VM), Vastus Lateralis (VL), Rectus Femoris (RF)
  Interventions: Other: Cura Kinesio-taping
- Placebo kinesio-taping (Placebo Comparator): consisted of 25 subjects who will receive placebo kinesio-taping across quadriceps.
  Interventions: Other: Placebo kinesio-taping

INTERVENTIONS:
Other: Cura Kinesio-taping — Cura tapes, a cotton strip with an acrylic adhesive. allows for unidirectional elasticity up to 60% beyond its resting length will be applied on origin to insertion on the superficial muscles of Quadriceps femoris (QF) (Vastus Medialis (VM), Vastus Lateralis (VL), Rectus Femoris (RF)
  Arms: Cura kinesio-taping
Other: Placebo kinesio-taping — Placebo kinesiotaping
  Arms: Placebo kinesio-taping

SUMMARY:
A Pretest post-test control group design will be used to investigate the effect of kinesio taping on electrical activity and peak torque of the quadriceps femoris muscle during concentric and eccentric contraction after arthroscopic partial meniscectomy (APM) surgery.

DETAILED DESCRIPTION:
Fifty patients after APM of any knee of both sexes will participate in this study after signing a written informed consent form approved.

from the ethical committee of Jazan University. They are selected according to the following Inclusion criteria:

1. All performed APM only without any other knee injury.
2. Finished the period of hospital stay (6-8 weeks)
3. Their age ranged from 20-40.
4. Their Body mass index ranged from 20-24.9 kg/m². 2- The subjects will be excluded from the study if they had one of th e following exclusion criteria: a- Knee or quadriceps disorders preventing physical stress. b- Subjects with cardiovascular or neurological problems. c- Smokers. d- Heavy caffeine intake subjects. 3- The subjects will be randomly assigned into two groups of equal numbers. Group A (Study) consisted of 66 subjects who will receive kinesio-taping from origin to insertion on the superficial muscles of the Quadriceps femoris (QF) (Vastus Medialis (VM), Vastus Lateralis (VL), Rectus Femoris (RF)). - Group B (Control) consisted of 66 subjects who will receive a placebo kinesio-taping across quadriceps. Anthropometric measures including "weight and height" and body. mass index (BMI) will be measured for all subjects in the first meeting before starting the evaluative procedures. All subjects were asked to shave the hair of their thigh before starting the evaluative procedure using blades, which was essential to prevent artifact during EMG evaluation and to facilitate the adherence of the tape to the skin. Bioelectrical activity and peak torque of quadriceps muscle of the lower extremity that had APM will be measured. The evaluation will be carried out before tapping, and then after the application of tapping for 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis only with arthroscopic partial meniscectomy
2. Must be finished a period of hospital stay (6-8 weeks)
3. Must have body mass index ranged from 20-24.9 kg/m².

Exclusion Criteria:

a. Knee or quadriceps disorders preventing physical stress. b- Cardiovascular or neurological problems. c- Smokers d- Heavy caffeine intake subjects.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Peak muscle torque | 1. Baseline: before tapping 2. after10 minutes of Cura kinesio-taping.
  Peak torque of the quadriceps femoris muscle during concentric and eccentric contraction after arthroscopic partial meniscectomy (APM) surgery using Biodex system
Bioelectrical activity of quadriceps muscle | 1. Baseline: before tapping 2. after10 minutes of Cura kinesio-taping.
  bioelectrical activity of the three quadriceps muscle heads will be measured. All subjects were asked to shave the hair of their thigh before starting.
  the evaluative procedure using blades, which was essential to prevent artifact during EMG evaluation and to facilitate the adherence of the tape to the skin

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Ahmed, Principal Investigator — Assistant Professor, Jazan University
Locations (1):
- Jazan University, Jizan, Gizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
I will share the data on request.